CLINICAL TRIAL: NCT04557189
Title: A Randomized Double-Blind, Sponsor-Open, Double-Dummy, Proof of Concept Phase 2 Study to Evaluate the Efficacy and Safety of TAK-951 Versus Ondansetron in the Prophylaxis of Postoperative Nausea and Vomiting in High-Risk Subjects
Brief Title: A Study of TAK-951 to Stop Adults Getting Nausea and Vomiting After Planned Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TAK-951-2001
Record Dates: First submitted 2020-09-18; First posted 2020-09-21 (Actual); Results first posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Postoperative Nausea and Vomiting (PONV)
Keywords: Drug Therapy
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ondansetron 4 mg IV (Experimental): Participants received prophylaxis with ondansetron 4 mg, intravenously (IV) immediately before induction and TAK-951 placebo subcutaneously (SC) approximately 30 to 45 minutes before the end of surgery (wound closure).
  Interventions: Drug: Ondansetron; Drug: TAK-951 Placebo
- TAK-951 4 mg SC (Experimental): Participants received prophylaxis with ondansetron placebo IV immediately before induction and TAK 951 4 mg, SC, approximately 30 to 45 minutes before the end of surgery (wound closure).
  Interventions: Drug: TAK-951; Drug: Ondansetron Placebo

INTERVENTIONS:
Drug: TAK-951 — TAK-951 SC injection
  Arms: TAK-951 4 mg SC
Drug: Ondansetron — Ondansetron IV injection
  Arms: Ondansetron 4 mg IV
Drug: Ondansetron Placebo — Ondansetron placebo-matching IV injection
  Arms: TAK-951 4 mg SC
Drug: TAK-951 Placebo — TAK-951 placebo-matching SC injection
  Arms: Ondansetron 4 mg IV

SUMMARY:
Some adults are at a higher risk of feeling sick (nausea) or being sick (vomiting) after they have surgery. In this study, these adults will have planned surgery. The main aim of this study is to learn if TAK-951 stops these adults from getting nausea or vomiting after surgery. This will be compared with another medicine called ondansetron. Another aim is to check for side effects from the study medicines.

Before surgery, the study doctor will check who can take part in this study. Those who can take part will be picked for either Treatment Group A or Treatment Group B by chance.

* Treatment Group A: Just before surgery, participants will receive a placebo slowly through a vein (infusion). Just before the end of the surgery, they will receive TAK-951 as an injection under the skin.
* Treatment Group B: Just before surgery, participants will receive ondansetron slowly through a vein (infusion). Just before the end of the surgery, they will receive a placebo as an injection under the skin. In this study, a placebo will look like TAK-951 but will not have any medicine in it.

Participants will not know which study medicines they received, or in which order, nor will their study doctors or surgeons. This is to help make sure the results are more reliable.

Participants will stay in the hospital for 24 hours after their surgery so that the study doctors can check for nausea and vomiting. The study doctors will also check for side effects from the study medicines.

Participants will visit the hospital for a check-up 14 days later.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-951. TAK-951 is being tested for prophylaxis for postoperative nausea and vomiting in high-risk participants.

The study will enroll a maximum of 160 patients, to allow a sample size of up to approximately 100 participants who have received both doses of Double-blind study drug/matching placebo. Participants will be randomly assigned in a 1:1 ratio to either Treatment Group A or Treatment Group B which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* Treatment Group A: Just before surgery, participants will receive a placebo slowly through a vein (infusion). Just before the end of the surgery, they will receive TAK-951 as an injection under the skin.
* Treatment Group B: Just before surgery, participants will receive ondansetron slowly through a vein (infusion). Just before the end of the surgery, they will receive a placebo as an injection under the skin. In this study, a placebo will look like TAK-951 but will not have any medicine in it.

This trial will be conducted in the United States. The overall time to participate in the study from the time of surgery to completion is approximately 14 days. Participants will make multiple visits to the clinic and will be contacted by telephone after receiving their last dose of the drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Participants undergoing elective surgery under general anesthesia, expected to last for at least 1 hour from induction of anesthesia to wound closure.
2. Participants are expected to require or have agreed to stay, at least 1 overnight in the hospital.
3. Participants American Society of Anesthesiologists (ASA) physical status is ASA I-III.
4. Participants with 3 or more Apfel risk factors defined as:

   1. Female sex.
   2. Nonsmoking status (never smoked or stopped smoking ≥12 months ago).
   3. History of PONV or motion sickness.
   4. Planned use of postoperative opioid analgesics.

Exclusion Criteria:

1. Participants who are expected to remain intubated post-anesthesia.
2. Participants who experience nausea or vomiting within 24 hours before surgery or are diagnosed with gastroparesis, cyclic vomiting syndrome, or other condition associated with acute or chronic nausea and vomiting.
3. Participants who have received, or are expected to receive, any excluded drug preoperatively within 24 hours before induction, during surgery, or within 24 hours after surgery.
4. Participants scheduled to receive neuraxial anesthesia (e.g., epidural, spinal, or caudal anesthesia), regional blocks, or total IV anesthesia, and/or planned to receive different drugs for premedication, induction, maintenance, or reversal of anesthesia than those specified in the protocol.
5. Participants who have an allergy or contraindication to the recommended and available rescue therapy for the treatment of PONV.
6. Circumstance that, in the investigator's opinion, make participation in this clinical study inappropriate.
7. Participants found at the screening to have a QT interval with Fridericia correction method (QTcF) ≥450 msec or other factors that increase the risk of QT prolongation or arrhythmic events. Assessments showing bundle branch block and a prolonged QTcF should be discussed with the study monitor and the sponsor for potential inclusion.
8. Participants who have a direct family history of premature sudden death or channelopathy, personal history of Brugada syndrome (right bundle branch block pattern with ST elevation in leads V1-V3), long QT, short QT, arrhythmogenic right ventricular dysplasia, hypertrophic cardiomyopathy or catecholaminergic polymorphic ventricular tachycardia (VT).
9. Participants who have had 3 incidents of vasovagal syncope within the last 5 years.
10. Participants with an average heart rate (HR) <55 or >100 bpm or systolic blood pressure (SBP) <90 mm Hg or Diastolic blood pressure (DBP) <60 mm Hg during screening or prior to randomization on the day of surgery.
11. Participants with a clinically significant ECG abnormality indicative of acute cardiac instability as determined by the investigator at screening, including more than first-degree atrioventricular block, nonsustained or sustained VT, or ECG changes consistent with acute myocardial ischemia or infarction.
12. Participants with a history of acute myocardial ischemia within the last 12 months.
13. Participants receiving beta-blockers chronically or between screening and surgery that cannot be safely withheld on the day of surgery in the investigator's judgment. Participants receiving certain other cardiovascular medications, such as vasodilators for hypertension, chronically or between screening and surgery that in the investigator's judgment cannot be adequately managed in the perioperative setting considering the potential vasodilatory effects of TAK-951 and anesthesia standard of care. The investigators must consult with the medical monitor regarding the eligibility of participants who are receiving beta-blockers, vasodilators, and other classes of medications that act on HR or BP.
14. Participants with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 times the upper limit of normal (ULN) or total bilirubin >1.5 times the ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (7):
- United States (7):
  - Helen Keller Hospital, Sheffield, Alabama
  - Lotus Clinical Research Inc, Pasadena, California
  - Phoenix Clinical Research, Tamarac, Florida
  - Stony Brook Medicine - Hospital, Stony Brook, New York
  - First Street Hospital - Research, Bellaire, Texas
  - Legent Orthopedic Hospital, Carrollton, Texas
  - Altus Houston Hospital - Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f94607b296beb001e63bf90

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 7 sites in the United States from 20 October 2020 to 21 March 2022. Participants with a diagnosis of postoperative nausea and vomiting (PONV) were enrolled in 1:1 ratio.
Pre-assignment Details: Participants received prophylaxis either with ondansetron before induction followed by TAK-951 placebo or prophylaxis with ondansetron placebo before induction followed by TAK-951 4 mg. Due to dosing error, of the 39 participants in the TAK-951 4 mg SC group, 18 participants received an unintended mis-dose of TAK-951 redacted mg. Data for these participants were collected and reported separately only for the outcome measures reporting data for the safety, pharmacokinetic, and immunogenicity set.
Period: Overall Study
Arm/Group | Ondansetron 4 mg IV | TAK-951 4 mg SC
Started | 44 | 45
Full Analysis Set (FAS) (FAS included all participants who were randomized to treatment and received both doses of double-blind study drug before and during surgery.) | 41 | 39
Pharmacokinetic (PK) Set (PK Set included all participants who received study drug and had at least 1 evaluable PK sample. Due to dosing error, an unintended mis-dose of TAK-951 redacted mg was administered to 18 participants from the TAK-951 4 mg group. Data for these participants were collected and reported separately.) | 0 | 21
Immunogenicity Set (Immunogenicity Set included all participants who received at least 1 dose of study drug, had an ADA status assessment at baseline, and at least 1 postbaseline sample. Due to dosing error, an unintended mis-dose of TAK-951 redacted mg was administered to 18 participants from the TAK-951 4 mg group. Data for these participants were collected and reported separately.) | 0 | 21
Unintended Mis-dose Due to Dosing Error (Of the 39 participants in the TAK-951 4 mg SC group, 18 participants received an unintended mis-dose of TAK-951 redacted mg.) | 0 | 18
Completed | 38 | 36
Not Completed | 6 | 9
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Reason not Specified | 3 | 6

BASELINE CHARACTERISTICS:
Population: FAS included all participants who were randomized to treatment and received both doses of double-blind study drug before and during surgery.
Groups:
- Ondansetron 4 mg IV: Participants received prophylaxis with ondansetron 4 mg, IV immediately before induction and TAK-951 placebo SC approximately 30 to 45 minutes before the end of surgery (wound closure).
- Total: Total of all reporting groups
Arm/Group | Ondansetron 4 mg IV | TAK-951 4 mg SC | Total
Number analyzed (Participants) | 41 | 39 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (10.32) | 45.1 (10.57) | 45.6 (10.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 38 | 76
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 17
  Not Hispanic or Latino | 33 | 29 | 62
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 10 | 18
  White | 31 | 27 | 58
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41 | 39 | 80
Weight [Mean (Standard Deviation); unit: kg] | 93.85 (27.439) | 87.61 (22.258) | 90.81 (25.087)
Height [Mean (Standard Deviation); unit: cm] | 164.57 (8.448) | 164.32 (9.499) | 164.44 (8.919)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI= Weight [kg]/Height [m]^2
  kg/m^2 | 34.41 (8.909) | 32.47 (7.574) | 33.47 (8.290)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response in the Immediate Postoperative Period
Description: Percentage of participants with complete response, defined as no emesis (vomiting or retching) and no need for rescue therapy (indicated if vomiting/retching and/or nausea score ≥4 or upon participant's request) were reported. The severity of nausea was scored using a self-reported, 11-point numerical Verbal Rating Scale (VRS), where 0 represents no nausea and 10 represents the worst nausea possible. Significant nausea was defined as a VRS score ≥4. Percentages are rounded off to whole number at the nearest single decimal.
Time Frame: 6 hours post-surgery (Day 1)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Ondansetron 4 mg IV | TAK-951 4 mg SC
Number analyzed (Participants) | 41 | 39
percentage of participants | 48.8 [0.335 to 0.641] | 71.8 [0.577 to 0.859]
Statistical Analysis 1: Comparison: Ondansetron 4 mg IV vs TAK-951 4 mg SC; Test type: Superiority; Adjusted Treatment Difference = 0.241, 95% CI 2-sided [0.031 to 0.452] — Adjusted treatment difference between TAK-951, ondansetron, associated confidence intervals: based on CMH method, adjusting for number of Apfel risk factors (3/4), or exact unconditional confidence limits for treatment difference if numerator is ≤5

2. Secondary Outcome: Percentage of Participants With Complete Response Within 24 Hours Post-Surgery
Description: as for outcome 1
Time Frame: Within 24 hours post-surgery (up to Day 2)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Ondansetron 4 mg IV | TAK-951 4 mg SC
Number analyzed (Participants) | 41 | 39
percentage of participants | 41.5 [0.264 to 0.565] | 59.0 [0.435 to 0.744]
Statistical Analysis 1: Comparison: Ondansetron 4 mg IV vs TAK-951 4 mg SC; Test type: Superiority; Adjusted Treatment Difference = 0.175, 95% CI 2-sided [-0.044 to 0.394]; Adjusted treatment difference between TAK-951, ondansetron, associated confidence intervals: based on Cochran-Mantel-Haenszel (CMH) method, adjusting for number of Apfel risk factors (3/4), or exact unconditional confidence limits for treatment difference if numerator is ≤5

3. Secondary Outcome: Percentage of Participants With Emesis in the First 6 Hours Post-Surgery
Description: Percentage of participants with emesis, defined as vomiting (the forceful discharge of even the smallest amount of stomach contents) or retching (the same muscular movements as vomiting but without expulsion of stomach contents) were reported. Percentages are rounded off to whole number at the nearest single decimal.
Time Frame: Within 6 hours post-surgery (Day 1)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Ondansetron 4 mg IV | TAK-951 4 mg SC
Number analyzed (Participants) | 41 | 39
percentage of participants | 17.1 [0.056 to 0.286] | 7.7 [0.016 to 0.209]
Statistical Analysis 1: Comparison: Ondansetron 4 mg IV vs TAK-951 4 mg SC; Test type: Superiority; Adjusted Treatment Difference = -0.094, 95% CI 2-sided [-0.253 to 0.059] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Participants With Emesis Within 24 Hours Post-Surgery
Description: as for outcome 3
Time Frame: Within 24 hours post-surgery (up to Day 2)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Ondansetron 4 mg IV | TAK-951 4 mg SC
Number analyzed (Participants) | 41 | 39
percentage of participants | 24.4 [0.112 to 0.375] | 10.3 [0.029 to 0.242]
Statistical Analysis 1: Comparison: Ondansetron 4 mg IV vs TAK-951 4 mg SC; Test type: Superiority; Adjusted Treatment Difference = -0.141, 95% CI 2-sided [-0.316 to 0.033] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Participants With Absence of Nausea in the First 6 Hours Post-Surgery
Description: Percentage of participants without nausea, defined as urge to vomit without the presence of expulsive muscular movements were reported. Percentages are rounded off to whole number at the nearest single decimal.
Time Frame: Within 6 hours post-surgery (Day 1)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Ondansetron 4 mg IV | TAK-951 4 mg SC
Number analyzed (Participants) | 41 | 39
percentage of participants | 41.5 [0.264 to 0.565] | 59.0 [0.435 to 0.744]
Statistical Analysis 1: Comparison: Ondansetron 4 mg IV vs TAK-951 4 mg SC; Test type: Superiority; Adjusted Treatment Difference = 0.191, 95% CI 2-sided [-0.029 to 0.410] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Percentage of Participants With Absence of Nausea in the First 24 Hours Post-Surgery
Description: Percentage of participants without nausea, defined as urge to vomit without the presence of expulsive muscular movements were reported. CMH method was used for analysis. Percentages are rounded off to whole number at the nearest single decimal.
Time Frame: Within 24 hours post-surgery (up to Day 2)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Ondansetron 4 mg IV | TAK-951 4 mg SC
Number analyzed (Participants) | 41 | 39
percentage of participants | 34.1 [0.196 to 0.487] | 48.7 [0.330 to 0.644]
Statistical Analysis 1: Comparison: Ondansetron 4 mg IV vs TAK-951 4 mg SC; Test type: Superiority; Adjusted Treatment Difference = 0.146, 95% CI 2-sided [-0.073 to 0.365] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Percentage of Participants Requiring Rescue Therapy for Breakthrough PONV Within 24 Hours Post-Surgery
Description: Percentage of participants to whom rescue therapy was given as per local standard of care guidelines were reported. Percentages are rounded off to whole number at the nearest single decimal.
Time Frame: Within 24 hours post-surgery (up to Day 2)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Ondansetron 4 mg IV | TAK-951 4 mg SC
Number analyzed (Participants) | 41 | 39
percentage of participants | 56.1 [0.409 to 0.713] | 33.3 [0.185 to 0.481]
Statistical Analysis 1: Comparison: Ondansetron 4 mg IV vs TAK-951 4 mg SC; Test type: Superiority; Adjusted Treatment Difference = -0.234, 95% CI 2-sided [-0.448 to -0.019] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Time From End of Surgery to First Emetic Event
Description: Duration between end of wound closure to first emetic event i.e., vomiting or retching was reported. If a participant did not have an emetic event within 24 hours post-surgery, they were censored at 24 hours post-surgery. Cox proportional hazard model was used for analysis.
Time Frame: Within 24 hours post-surgery (up to Day 2)
Population: FAS included all participants who were randomized to treatment and received both doses of double-blind study drug before and during surgery. Overall number analyzed are the number of participants with events.
Measure: Median (Full Range); unit: hours
Arm/Group | Ondansetron 4 mg IV | TAK-951 4 mg SC
Number analyzed (Participants) | 10 | 4
hours | NA [NA to NA] — Median time to first event and full range are not estimable due to too few events within the 24 hours observation window. | NA [NA to NA] — Median time to first event and full range are not estimable due to too few events within the 24 hours observation window.
Statistical Analysis 1: Comparison: Ondansetron 4 mg IV vs TAK-951 4 mg SC; Test type: Superiority; Hazard Ratio (HR) = 0.393, 95% CI 2-sided [0.122 to 1.259] — The hazard ratio is derived from a Cox proportional hazard model with treatment group and the number of Apfel risk factors (3 or 4) as independent variables

9. Secondary Outcome: Peak Nausea Verbal Rating Scale (VRS) Score
Description: VRS was used to score postoperative nausea on 11-point numerical scale. The score ranges from 0-10, where 0 represents 'no nausea' and 10 represents 'worst nausea possible'. Higher score represents worsening of disease. Mixed-effects model for repeated measures (MMRM) was used for analysis. Least square mean (LSM) estimates extracted from MMRM are presented in the data table for each time point.
Time Frame: 30 minutes; 1, 2, 6, and 24 hours post-surgery (up to Day 2)
Population: FAS included all participants who were randomized to treatment and received both doses of double-blind study drug before and during surgery. Overall number of participants analyzed are the participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ondansetron 4 mg IV | TAK-951 4 mg SC
Number analyzed (Participants) | 18 | 26
score on a scale
  30 Minutes Post Surgery: number analyzed (Participants) | 17 | 25
  30 Minutes Post Surgery | 0.159 (0.227) | 0.347 (0.184)
  1 Hour Post Surgery: number analyzed (Participants) | 17 | 26
  1 Hour Post Surgery | 0.099 (0.254) | 0.500 (0.204)
  2 Hours Post Surgery: number analyzed (Participants) | 17 | 26
  2 Hours Post Surgery | 0.043 (0.201) | 0.308 (0.162)
  6 Hours Post Surgery | -0.020 (0.073) | 0.077 (0.059)
  24 Hours Post Surgery | 0.203 (0.142) | 0.000 (0.117)
Statistical Analysis 1: Comparison: Ondansetron 4 mg IV vs TAK-951 4 mg SC; 30 Minutes Post Surgery; Test type: Superiority; Difference in LSM Estimates = 0.188, 95% CI 2-sided [-0.402 to 0.777]; From MMRM analysis over all post-randomization timepoints, with the Peak VRS score as the outcome, treatment group, timepoint, number of Apfel risk factors and treatment-by-timepoint interaction as fixed effects and participant as random effect with unstructured covariance structure for observed data up to 24 hours post surgery
Statistical Analysis 2: Comparison: Ondansetron 4 mg IV vs TAK-951 4 mg SC; 1 Hour Post Surgery; Test type: Superiority; Difference in LSM Estimates = 0.401, 95% CI 2-sided [-0.258 to 1.059]; [other analysis details as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Ondansetron 4 mg IV vs TAK-951 4 mg SC; 2 Hours Post Surgery; Test type: Superiority; Difference in LSM Estimates = 0.265, 95% CI 2-sided [0 to 0.786]; [other analysis details as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Ondansetron 4 mg IV vs TAK-951 4 mg SC; 6 Hours Post Surgery; Test type: Superiority; Difference in LSM Estimates = 0.097, 95% CI 2-sided [-0.093 to 0.286]; [other analysis details as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: Ondansetron 4 mg IV vs TAK-951 4 mg SC; 24 Hours Post Surgery; Test type: Superiority; Difference in LSM Estimates = -0.203, 95% CI 2-sided [-0.575 to 0.170]; [other analysis details as in outcome 9, analysis 1]

10. Secondary Outcome: Percentage of Participants With Total Response
Description: Percentage of participants with total response, defined as no emesis, no nausea (VRS score <1), and no need for rescue therapy were reported. VRS was used to score postoperative nausea on 11-point numerical scale, where 0 represents 'no nausea' and 10 represents 'worst nausea possible'. Percentages are rounded off to whole number at the nearest single decimal.
Time Frame: Within 24 hours post-surgery (up to Day 2)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Ondansetron 4 mg IV | TAK-951 4 mg SC
Number analyzed (Participants) | 41 | 39
percentage of participants | 34.1 [0.196 to 0.487] | 48.7 [0.330 to 0.644]
Statistical Analysis 1: Comparison: Ondansetron 4 mg IV vs TAK-951 4 mg SC; Test type: Superiority; Adjusted Treatment Difference = 0.146, 95% CI 2-sided [-0.073 to 0.365] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: TAK-951 Plasma Concentrations
Time Frame: 1-3, 4-6, 7-9, 10-18, and 22-26 hours post-dose (up to Day 2)
Population: PK Set included all participants who received study drug and had at least 1 evaluable PK sample. Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analysis at the specified timepoint. The data for this outcome measure was collected and reported separately for the participants who received the unintended mis-dose of TAK-951 redacted mg.
Measure: Mean (Standard Deviation); unit: picograms per milliliter(pg/mL)
Groups:
- TAK-951 Redacted mg SC: Participants received prophylaxis with ondansetron placebo IV immediately before induction and unintended mis-dose of TAK 951 redacted mg, SC, approximately 30 to 45 minutes before the end of surgery (wound closure).
Arm/Group | TAK-951 4 mg SC | TAK-951 Redacted mg SC
Number analyzed (Participants) | 20 | 18
picograms per milliliter(pg/mL)
  1-3 Hours Post Dose: number analyzed (Participants) | 20 | 17
  1-3 Hours Post Dose | 24734.50 (14782.359) | 58229.41 (42971.281)
  4-6 Hours Post Dose: number analyzed (Participants) | 18 | 18
  4-6 Hours Post Dose | 18456.11 (13906.450) | 36950.00 (26649.650)
  7-9 Hours Post Dose: number analyzed (Participants) | 16 | 17
  7-9 Hours Post Dose | 10568.31 (8140.684) | 17741.76 (9705.848)
  10-18 Hours Post Dose: number analyzed (Participants) | 9 | 0
  10-18 Hours Post Dose | 4478.22 (2433.185) |
  22-26 Hours Post Dose: number analyzed (Participants) | 10 | 0
  22-26 Hours Post Dose | 672.63 (699.161) |

12. Secondary Outcome: Percentage of Participants With Any Treatment Emergent Adverse Event (TEAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE is defined as an AE with an onset that occurs after receiving study drug. Percentages are rounded off to whole number at the nearest single decimal.
Time Frame: From first administration of study drug up to Day 14
Population: Safety Analysis Set (SAF) included all participants who were randomized to treatment and received both doses of double-blind study drug. The data for this outcome measure was collected and reported separately for the participants who received the unintended mis-dose of TAK-951 redacted mg.
Measure: Number; unit: percentage of participants
Arm/Group | Ondansetron 4 mg IV | TAK-951 4 mg SC | TAK-951 Redacted mg SC
Number analyzed (Participants) | 41 | 21 | 18
percentage of participants | 87.8 | 71.4 | 88.9

13. Secondary Outcome: Percentage of Participants With Markedly Abnormal Vital Signs
Description: Vital signs included heart rate, respiratory rate, systolic blood pressure (SBP) and diastolic blood pressure (DBP), body temperature and BMI. Percentage of participants with markedly abnormal vital sign values were reported. Percentages are rounded off to whole number at the nearest single decimal. Only categories with at least 1 participant with data are reported.
Time Frame: From first administration of study drug up to Day 14
Population: SAF included all participants who were randomized to treatment and received both doses of double-blind study drug. The data for this outcome measure was collected and reported separately for the participants who received the unintended mis-dose of TAK-951 redacted mg.
Measure: Number; unit: percentage of participants
Arm/Group | Ondansetron 4 mg IV | TAK-951 4 mg SC | TAK-951 Redacted mg SC
Number analyzed (Participants) | 41 | 21 | 18
percentage of participants
  Heart Rate (beats per minute [beats/min]): Low: <60 | 36.6 | 19.0 | 22.2
  Heart Rate (beats/min): High: >100 | 14.6 | 66.7 | 72.2
  Respiratory Rate (breaths per minute [breaths/min]): Low: <12 | 46.3 | 19.0 | 55.6
  Respiratory Rate (breaths/min): High: >16 | 100.0 | 100.0 | 100.0
  SBP (millimeters of mercury [mmHg]): Low: <85 | 7.3 | 9.5 | 16.7
  SBP (mmHg): High: >140 | 70.7 | 42.9 | 77.8
  DBP (mmHg): Low: <50 | 22.0 | 33.3 | 55.6
  DBP (mmHg): High: >90 | 43.9 | 14.3 | 38.9
  BMI (kg/m^2): High: >25.0 | 90.2 | 85.7 | 88.9

14. Secondary Outcome: Percentage of Participants With Clinically Significant Electrocardiogram (ECG)
Description: Percentage of participants with clinically significant ECG interpretation were reported. Percentages are rounded off to whole number at the nearest single decimal. A combined ECG interpretation was derived using ECG heart rate, PR interval, RR interval, QRS duration, QT interval, and QT interval with Fridericia correction method (QTcF).
Time Frame: From first administration of study drug up to Day 14
Population: SAF included all participants who were randomized to treatment and received both doses of double-blind study drug. The data for this outcome measure was collected and reported separately for the participants who received the unintended mis-dose of TAK-951 redacted mg. Overall number analyzed is the number of participants with data available for analyses. Clinical significance is based on PI determination.
Measure: Number; unit: percentage of participants
Arm/Group | Ondansetron 4 mg IV | TAK-951 4 mg SC | TAK-951 Redacted mg SC
Number analyzed (Participants) | 41 | 20 | 18
percentage of participants | 2.4 | 0.0 | 0.0

15. Secondary Outcome: Percentage of Participants With Markedly Abnormal Clinical Laboratory Values
Description: Laboratory parameters included hematology and serum chemistry. Percentage of participants with markedly abnormal clinical laboratory values were reported. Percentages are rounded off to whole number at the nearest single decimal. Only categories with at least 1 participant with data are reported.
Time Frame: From first administration of study drug up to Day 14
Population: SAF included all participants who were randomized to treatment and received both doses of double-blind study drug. Number analyzed is the number of participants with data available for analysis for the specified category. The data for this outcome measure was collected and reported separately for the participants who received the unintended mis-dose of TAK-951 redacted mg.
Measure: Number; unit: percentage of participants
Arm/Group | Ondansetron 4 mg IV | TAK-951 4 mg SC | TAK-951 Redacted mg SC
Number analyzed (Participants) | 41 | 21 | 18
percentage of participants
  Erythrocytes (10^12 per liter [10^12/L]): Low: <0.8*Lower Limit of Normal (LLN) | 14.6 | 14.3 | 27.8
  Hemoglobin (grams per liter [g/L]): Low: <0.8*LLN | 14.6 | 23.8 | 11.1
  Hematocrit (percent [%]): Low: <0.8*LLN | 12.2 | 23.8 | 11.1
  Aspartate Aminotransferase (units per liter[U/L]): High: >3*Upper Limit of Normal (ULN) | 0.0 | 4.8 | 0.0
  Alanine Aminotransferase (U/L): High: >3*ULN | 0.0 | 4.8 | 0.0
  Albumin (g/L): Low: <25 | 0.0 | 4.8 | 0.0
  Protein (g/L): Low: <0.8*LLN | 2.4 | 4.8 | 16.7
  Gamma Glutamyl Transferase (U/L): High: >3*ULN: number analyzed (Participants) | 41 | 20 | 18
  Gamma Glutamyl Transferase (U/L): High: >3*ULN | 0.0 | 5.0 | 0.0
  Glucose (millimoles per liter [mmol/L]): Low: <3 | 0.0 | 4.8 | 0.0
  Glucose (millimoles per liter [mmol/L]): High: >10 | 4.9 | 0.0 | 0.0
  Potassium (mmol/L): High: >5.5 | 2.4 | 0.0 | 0.0

16. Secondary Outcome: Percentage of Participants With TAK-951 Antidrug Antibodies (ADA)
Description: Percentage of participants with ADA results as: ADA negative, ADA positive were reported. Participants with ADA positive status are defined as those who had confirmed positive ADA status in baseline or at least 1 postbaseline assessments. Participants with ADA negative status are defined as those who did not have positive ADA response at baseline and in all postbaseline assessments.
Time Frame: Within 6 hours post-surgery (Day 1)
Population: Immunogenicity Set included all participants who received at least 1 dose of study drug, had an ADA status assessment at baseline, and at least 1 postbaseline sample. Overall number analyzed is the number of participants with non-missing data for this outcome measure i.e., responders. The data for this outcome measure was collected and reported separately for the participants who received the unintended mis-dose of TAK-951 redacted mg.
Measure: Number; unit: percentage of participants
Arm/Group | TAK-951 4 mg SC | TAK-951 Redacted mg SC
Number analyzed (Participants) | 14 | 14
percentage of participants
  Any Antidrug Antibody Positive | 0.0 | 0.0
  Any Antidrug Antibody Negative | 100.0 | 100.0

ADVERSE EVENTS:
Time Frame: From first administration of study drug up to Day 14
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. FAS included all participants who were randomized to treatment and received both doses of double-blind study drug before and during surgery. The data is reported per dose received by participants.
Arm/Group | Ondansetron 4 mg IV | TAK-951 4 mg SC | TAK-951 Redacted mg SC
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/21 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/21 | 0/18
Other Adverse Events (participants affected / at risk) | 36/41 | 15/21 | 16/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ondansetron 4 mg IV (N=41) | TAK-951 4 mg SC (N=21) | TAK-951 Redacted mg SC (N=18)
Bradycardia (Cardiac disorders) | 4 | 0 | 0
Chills (General disorders) | 1 | 2 | 0
Flatulence (Gastrointestinal disorders) | 6 | 6 | 1
Hypertension (Vascular disorders) | 1 | 0 | 2
Hypotension (Vascular disorders) | 3 | 1 | 7
Procedural hypotension (Injury, poisoning and procedural complications) | 16 | 8 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 4 | 6 | 10
Tachycardia (Cardiac disorders) | 0 | 0 | 3
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 4
Anxiety (Psychiatric disorders) | 1 | 0 | 1
Blood pressure increased (Investigations) | 1 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/89/NCT04557189/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/89/NCT04557189/SAP_001.pdf